CLINICAL TRIAL: NCT00517569
Title: Phase I Study for Assessment of Safety of Gene Therapy With GX-12 in Combination With HAART for the HIV-1 Infected Patients
Brief Title: Gene Therapy With GX-12 in Combination With HAART for the HIV-1 Infected Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genexine, Inc. (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Prof. Kang-Won Choe / Principal Investigator, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GX-12_HIV_I
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections
Keywords: Gene Therapy; GX-12; HIV-1; Interleukin; AIDS; HIV-1 type B infection; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): GX-12 combined with HAART
  Interventions: Genetic: GX-12; Drug: HAART

INTERVENTIONS:
Genetic: GX-12 — a mixed plasma DNA (HIV-1 antigen genes and human IL-12 mutant) 4, 8, 16mg, i.m., once every other weeks for 22 weeks (total 12 times)
Drug: HAART — Highly active antiretroviral therapy; Discontinuation at 24 weeks; NB: The patients should be treated with 2 NRTIs+1 NNRTI or 2 NRTIs + 1 PI, according to the guidelines published by DHHS in the USA.

SUMMARY:
The purpose of this study is to assess the safety of GX-12 gene therapy combined with HAART in the HIV-1 infected patients and to investigate the efficacy with the value of plasma viral load and with CD4 counts and HIV-1 specific IFN-gamma expressed T-lymphocytes

DETAILED DESCRIPTION:
Currently, management of HIV infection and AIDS is mainly done by antiviral chemotherapy which inhibits reverse transcriptase or proteolytic enzyme. The HAART (highly active antiretroviral therapy) has indeed succeeded extraordinary in decrease of the mortality and in increase of the life expediency of AIDS patients. However, there have been some significant limitations of them (for example, treatment fatigues, the side effects, the emergency of resistant, high medical costs, etc.).

Recently, there has been a number of bioresearch for immunotherapy to overcome these limitations of current medications. GX-12 is a genetic using a naked DNA with human IL-12 mutant as immune adjuvant. GX-12 is designed to vaccinate the individuals with HIV antigens, which is to result in enhancing the HIV specific immunity and to expand broadly the immune responses nonspecifically.

In this study, the safety and efficacy of GX-12 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50 years
* HIV-1 type B infected but asymptomatic patient
* Patient who has received HAART less than 6 months according to the standard management guidelines and reached to aviremia
* Patient with appropriate immunity (i.e., CD4 counts>=400cells/ul and SI>3 by CD4+ T-cell proliferation in vitro assay)
* Patient with negative HBV and HCV
* Woman who is not childbearing or who has used any contraceptive at least for 3 months before study entry
* Patients given a written consent

Exclusion Criteria:

* Patient who has received other investigational drug or who participated into other study within 30 days before this study
* Patient who had an experience of hypersensitivity to same drug (for example: a plasmid DNA, etc)
* Patient who has received an immunosuppressant
* Patient who has received other HIV vaccine
* Patient who has received other interleukin(s)
* Patient who experienced an opportunistic infection defined as AIDS before this study
* Patient with any severe recurrent diarrhea or vomiting
* Patient with clinically significant acute or chronic liver dysfunction, kidney dysfunction, hematological disorder, endocrine disorder, immune disorder, heart disease, infection, etc.
* Patient with malignant tumor(s)
* Patient with alcohol or drug abuse
* Patient of potential harm due to drug interactions by HAART
* Woman of pregnancy (positive pregnancy test) or beast feeding
* Patient who is not appropriate at investigator's discretion, not specified in above

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Safety: adverse events and laboratory abnormalities | 36 weeks

SECONDARY OUTCOMES:
Primary efficacy endpoint: plasma viral load Secondary efficacy endpoint: CD4 counts and HIV-1 Antigen specific IFN-gamma expressed T-lymphocytes | 24, 28, 32 and 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: KANG-WON CHOE, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea